CLINICAL TRIAL: NCT06479486
Title: Clinimetric Properties of Performance-based Measures of Physical Function in Patients With COPD: a Comparison of Clinimetric Properties of Four Tools
Brief Title: Clinimetric Properties of Performance-based Measures of Physical Function in Patients With COPD
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aimen Shahbaz
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Clinimetric properties, COPD, performance-based measures
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functionality Assessment (Other): Each participant will be provided with an informed consent form detailing the purpose of the study. After obtaining written consent, baseline data will be collected, including demographic information, medical history, and any pre-existing conditions.The participants will then undergo the post-laparotomy interventions as described. Throughout the intervention period, data will be collected using the tools mentioned: 6 minute Walk Test, 30 seconds sit to stand test, 2 Minute walk Test, and Timed Up and GO to determine any changes in their functionality test .For reliability, test retest will be conducted both on day 1 and on the next day.
  Interventions: Diagnostic Test: Assigned Interventions

INTERVENTIONS:
Diagnostic Test: Assigned Interventions — warm up: global range of motion exercises; breathing control. Aerobic training: walking, cycling, stepping Resistance training: free weights(major muscle groups of upper and lower limbs and trunk Cool down; Breathing control and stretching exercises.
  Other Names: Standardized pulmonary rehab protocols

SUMMARY:
A COPD (Chronic obstructive pulmonary disease), is a group of progressive lung diseases. COPD is a preventable and treatable respiratory disorder largely caused by smoking and long term exposure to chemical irritants. This study aims to provide essential insights into the reliability, validity, responsiveness and Interpretability of such tests, enabling healthcare professionals to make informed decisions about patient recovery progress and the optimization of rehabilitation protocols.

DETAILED DESCRIPTION:
A COPD (Chronic obstructive pulmonary disease), is a group of progressive lung diseases, a preventable and treatable respiratory disorder largely caused by smoking and long term exposure to chemical irritants. COPD affects the respiratory system and is progressive, which can result in a number of difficulties or impairments. ) Effect on Daily Activities, Work Limitations, Fatigue Muscle Weakness, Breathlessness and Reduced Exercise Capacity, and Impaired Quality of Life. Pulmonary rehabilitation is a comprehensive course that helps people with chronic respiratory illnesses, such as COPD, improve their overall health and quality of life. Clinimetric properties of four distinct tools designed for assessing performance-based physical functional outcomes following COPD patients surgery. 6 Minute Walk Test (6MWT), 2 minute Walk test (2MWT), and Timed Up and GO (TUG), 30sec sit to stand test (30sec STS) will be assessed to determine any changes in their functionality test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of COPD (FEV1/FVC < 0.70).
* Both genders
* Clinically stable
* Age 40-65 years

Exclusion Criteria:

* Disease exacerbation in last 4 weeks
* Co-existing respiratory or any other condition
* Inability to perform tests due to cognitive or any physical limitations

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
6MWT (Six-Minute Walk Test) | 6 week
  A six-minute walk test to assess your fitness or functional condition. Using a pulse oximeter, the researchers will take your blood pressure, pulse, and oxygen saturation before you start walking. The following instructions will be given to participants. The competitors will walk as close to a chair or cone as they can for six minutes at their regular pace. After that, they will turn around and continue walking back and forth for an additional six minutes. It was shown that this test had good test-retest reliability.
2MWT (Two-Minute Walk Test) | 6 week
  The 2MWT is a functional exercise test designed to evaluate an individual's aerobic capacity and endurance over a shorter duration compared to the 6MWT.
Timed Up and GO (TUG) | 6 week
  It is designed to assess an individual's mobility and requires the participant to stand up from a seated position, walk a distance of three meters, turn around, walk back to the chair, and sit down.
30 seconds sit to stand test (30SSTS): | 6 week
  Used to assess lower extremity strength, balance, and functional capacity in patients with chronic obstructive pulmonary disease (COPD). It involves measuring the number of times a patient can rise from a seated position to a full standing position and then return to sitting within a 30-second period. The test is typically conducted in a chair with a standardized height and armrest comapred TUG test

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Hearts International Hospital, Islamabad, AL, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Massierer D, Alsowayan W, Lima VP, Bourbeau J, Janaudis-Ferreira T. Prognostic value of simple measures of physical function and muscle strength in COPD: A systematic review. Respir Med. 2020 Jan;161:105856. doi: 10.1016/j.rmed.2019.105856. Epub 2019 Dec 19. PMID 32056729
- [Background] Charlson ME, Carrozzino D, Guidi J, Patierno C. Charlson Comorbidity Index: A Critical Review of Clinimetric Properties. Psychother Psychosom. 2022;91(1):8-35. doi: 10.1159/000521288. Epub 2022 Jan 6. PMID 34991091